CLINICAL TRIAL: NCT00921882
Title: Is it Possible to Screen for Type 2 Diabetes at Day 2 Gestational Diabetes Mellitus Postpartum?
Brief Title: Is it Possible to Screen for Type 2 Diabetes at Day 2 in Gestational Diabetes Mellitus Patients Postpartum?
Acronym: DG4
Status: Completed | Type: Observational
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Jean-Luc Ardilouze, Endocrinologist, researcher, Université de Sherbrooke
Other Study IDs: 07-084
Record Dates: First submitted 2009-06-10; First posted 2009-06-16 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Gestational Diabetes Mellitus; Type 2 Diabetes
Keywords: Type 2 diabetes; Post-partum screening
MeSH Terms: conditions — Diabetes, Gestational; Diabetes Mellitus, Type 2 | interventions — Glucose Tolerance Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Oral glucose tolerance test: oral glucose tolerance test performed 48 hours post-partum and 8 weeks post-partum.
  Interventions: Procedure: Oral glucose tolerance test

INTERVENTIONS:
Procedure: Oral glucose tolerance test — Subjects will have the Oral glucose tolerance test 48 hours post-partum and the same test 8 weeks post-partum.

SUMMARY:
Within 6 months of delivery, women who had gestational diabetes mellitus should be screened for type 2 diabetes with a fasting plasma glucose test and/or a 2-h postchallenge glycemia in a 75-g oral glucose tolerance test. However, not all women are screened. The objective of this study is to compare the screening test for type 2 diabetes done at 48 hours post-partum versus 8 weeks post-partum. The investigators want to measure the specificity, sensitivity, false and true predictive values of the screening test at 48 hours post-partum compared to the gold-standard.

ELIGIBILITY:
Inclusion Criteria:

* Dx of gestational diabetes treated with insulin
* To be in post-partum
* Delivery of a baby of at least 37 weeks of gestation
* Have signed the consent form

Exclusion Criteria:

* History of glucose intolerance of diabetes before the pregnancy
* Obstetrical pathology during pregnancy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women with gestational diabetes mellitus who delivered.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2008-06 (Actual); Primary Completion 2012-10 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Oral glucose tolerance test | 8 weeks post partum
  Sensitivity, specificity, true and false predictive values of the oral glucose tolerance test

SECONDARY OUTCOMES:
Acceptability of screening test | 8 weeks post partum
  Prefered moment to do the screening test (48 hours post partum or 8 weeks post partum)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc Ardilouze, MD, PhD, Principal Investigator — Université de Sherbrooke
Locations (1):
- Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec, Canada